CLINICAL TRIAL: NCT00310310
Title: Effect of Self-Management on Improving Sleep Apnea Outcomes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: IIR 02-275
Record Dates: First submitted 2006-03-30; First posted 2006-04-03 (Estimated); Results first posted 2017-03-22 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-03

CONDITIONS: Sleep Apnea Syndromes
Keywords: Continuous positive airway pressure; Patient compliance; Self-care
MeSH Terms: conditions — Sleep Apnea Syndromes; Patient Compliance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care (Placebo Comparator): Usual sleep apnea and cpap care
  Interventions: Behavioral: Usual care
- Self-Management (Experimental): sleep apnea self-management program - 4 sessions, group-based
  Interventions: Behavioral: Sleep Apnea Self-Management Program

INTERVENTIONS:
Behavioral: Sleep Apnea Self-Management Program — Sleep apnea self-management program - 4 sessions, group-based.
  Arms: Self-Management
Behavioral: Usual care — Usual sleep apnea and cpap care
  Arms: Usual Care

SUMMARY:
Obstructive sleep apnea syndrome (OSA) is a common sleep disorder that is associated with serious medical and psychological complications. Nasal continuous positive airway pressure (CPAP) is the treatment of choice for this condition because it is highly effective in reducing the frequency of nocturnal respiratory events, improving sleep architecture, decreasing daytime sleepiness and improving blood pressure. Incomplete patient adherence, however, limits the effectiveness of CPAP therapy and results in sub-optimal patient outcomes. Previous efforts to enhance CPAP adherence have resulted in only modest improvements, have generally not been theory-driven, and have had minimal effects on key patient outcomes such as reduction in OSA symptoms or increase in health-related quality of life (HRQOL). The planned intervention in this proposal, the Sleep Apnea Self-Management Program (SASMP), is based on the rationale that sleep apnea is a chronic disease that requires significant self-care on the part of the patient. We draw on the extensive chronic disease self-management literature to provide a solid theoretical justification for this pragmatic intervention both to better manage key aspects of OSA and to increase CPAP adherence. Chronic disease management programs help reduce symptoms, improve HRQOL, improve treatment adherence, and decrease medical utilization.

DETAILED DESCRIPTION:
Background: Obstructive sleep apnea syndrome (OSA) is a common sleep disorder that is associated with serious medical and psychological complications. Nasal continuous positive airway pressure (CPAP) is the treatment of choice for this condition because it is highly effective in reducing the frequency of nocturnal respiratory events, improving sleep architecture, decreasing daytime sleepiness and improving blood pressure. Incomplete patient adherence, however, limits the effectiveness of CPAP therapy and results in sub-optimal patient outcomes. Previous efforts to enhance CPAP adherence have resulted in only modest improvements, have generally not been theory-driven, and have had minimal effects on key patient outcomes such as reduction in OSA symptoms or increase in health-related quality of life (HRQOL). The planned intervention in this proposal, the Sleep Apnea Self-Management Program (SASMP), is based on the rationale that sleep apnea is a chronic disease that requires significant self-care on the part of the patient. We draw on the extensive chronic disease self-management literature to provide a solid theoretical justification for this pragmatic intervention both to better manage key aspects of OSA and to increase CPAP adherence. Chronic disease management programs help reduce symptoms, improve HRQOL, improve treatment adherence, and decrease medical utilization. Objectives: The primary aim of this study is to compare the efficacy of the SASMP to Usual Care for improving OSA symptom status, HRQOL, and self-reported medical utilization. A second aim is to examine the extent to which changes in symptoms and HRQOL are mediated by changes in self-efficacy and CPAP adherence. Methods: We will evaluate the Sleep Apnea Self-Management Program (SASMP) by conducting a randomized, controlled trial of the program compared to Usual Care in patients diagnosed with OSA and prescribed CPAP therapy. Participants randomized to the SASMP group will attend 4 weekly educational sessions of 2.5 hours each. Two trained leaders facilitate the program from a scripted manual. Key topics covered in this program include 1) management of OSA symptoms, CPAP side effects, and weight loss; 2) maintaining social contacts and family relationships; and 3) dealing with symptoms of depression and worries about the future. Findings: No results at this time. Status: We are currently engaging in start-up activities. Impact: The results of this project can improve service delivery and improve health outcomes for sleep apnea patients at the Veterans Affairs San Diego Healthcare System, throughout the VA, as well as to any community based sleep clinic.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of obstructive sleep apnea
* No previous use of CPAP
* Must be a Veteran with residence within San Diego County

Exclusion Criteria:

* Home oxygen therapy
* Fatal comorbidities (i.e., life expectancy less than 6 mos)
* Contraindications for CPAP use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2006-04; Primary Completion 2009-05 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl J Stepnowsky, PhD, Principal Investigator — San Diego Veterans Healthcare System
Locations (1):
- VA San Diego Healthcare System, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stepnowsky CJ, Palau JJ, Gifford AL, Ancoli-Israel S. A self-management approach to improving continuous positive airway pressure adherence and outcomes. Behav Sleep Med. 2007;5(2):131-46. doi: 10.1080/15402000701190622. PMID 17441783
- [Result] Stepnowsky CJ, Palau JJ, Marler MR, Gifford AL. Pilot randomized trial of the effect of wireless telemonitoring on compliance and treatment efficacy in obstructive sleep apnea. J Med Internet Res. 2007 May 17;9(2):e14. doi: 10.2196/jmir.9.2.e14. PMID 17513285
- [Result] Stepnowsky CJ, Ancoli-Israel S. Sleep and Its Disorders in Seniors. Sleep Med Clin. 2008;3(2):281-293. doi: 10.1016/j.jsmc.2008.01.011. No abstract available. PMID 19122865
- [Derived] Deering S, Liu L, Zamora T, Hamilton J, Stepnowsky C. CPAP Adherence is Associated With Attentional Improvements in a Group of Primarily Male Patients With Moderate to Severe OSA. J Clin Sleep Med. 2017 Dec 15;13(12):1423-1428. doi: 10.5664/jcsm.6838. PMID 29065955

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and screened from the Pulmonary Sleep/CPAP Clinic at the Veterans Affairs San Diego Healthcare System (VASDHS). Project offices were based at the VASDHS HSR&D unit.
Period: Overall Study
Arm/Group | Usual Care | Self-Management
Started | 120 | 120
Completed | 90 | 100
Not Completed | 30 | 20

BASELINE CHARACTERISTICS:
Population: The target population for this study is all Veterans with OSA. It was expected that most participants would be middle-aged and older men and women, from a variety of ethnic backgrounds and with a full range of medical co-morbidities.
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | Self-Management | Total
Number analyzed (Participants) | 120 | 120 | 240
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.1 (12.5) | 56.3 (11.9) | 56.2 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 116 | 118 | 234
Region of Enrollment [Number; unit: participants]
  United States | 120 | 120 | 240

OUTCOME MEASURES:

1. Primary Outcome: CPAP Adherence
Description: The investigators examined the data obtained in the Sleep Apnea Self-Management Program at the one-month time point relative to participation in the Usual Care group.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: hours per night
Arm/Group | Usual Care | Self-Management
Number analyzed (Participants) | 90 | 100
hours per night | 2.8 (2.6) | 3.9 (2.4)
Statistical Analysis 1: Comparison: Usual Care vs Self-Management; Test type: Superiority or Other; p = 0.001, t-test, 1 sided

2. Primary Outcome: CPAP Adherence
Description: The investigators also examined the data obtained at the 6-month time point.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: hours per night
Arm/Group | Usual Care | Self-Management
Number analyzed (Participants) | 90 | 100
hours per night | 2.3 (2.5) | 3.1 (2.5)
Statistical Analysis 1: Comparison: Usual Care vs Self-Management; Test type: Superiority or Other; p = 0.023, t-test, 1 sided

3. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire aimed at assessing sleep quality and disturbances over a 1-month period.79 The PSQI measures seven areas of sleep: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. Items are answered utilizing a Likert scale with 0 being indicative of better sleep and the maximum value of 3 being indicative of poor sleep. The PSQI has acceptable reliability (Cronbach's alpha = 0.83), test-retest reliability of 0.85, and can distinguish good and poor sleepers (global PSQI score > 5 has diagnostic sensitivity = 89.6% and specificity 86.5%).
  In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Time Frame: 1 Month
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Self-Management
Number analyzed (Participants) | 90 | 100
units on a scale | 8.5 (2.9) | 8.4 (3.2)
Statistical Analysis 1: Comparison: Usual Care vs Self-Management; Test type: Superiority or Other; p = 0.8, t-test, 1 sided

4. Secondary Outcome: Pittsburgh Sleep Quality Index (PSQI)
Description: as for outcome 3
Time Frame: 6 Months
Population: The target population for this study is all Veterans with OSA. It was expected that most participants would be middle-aged and older men and women, from a variety of ethnic backgrounds and with a full range of medical co-morbidities. We had a few Veterans who skipped this assessment when filling out the project assessment packet.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Self-Management
Number analyzed (Participants) | 78 | 89
units on a scale | 8.4 (3.6) | 8.3 (3.3)

5. Other Pre Specified Outcome: Sleep Apnea Quality of Life Index (SAQLI)
Description: Sleep Apnea Quality of Life Index (SAQLI) which is a 35-item clinician-administered scale composed of five domains: daily functioning, social interactions, emotional functioning, symptoms, and CPAP side effects. . It has high internal consistency, strong content and construct validity, and adequate concurrent and discriminative validity, and is responsive to changes in HRQOL. The key advantages to inclusion of the SAQLI is that it is the only clinician-administered scale in the study and it contains a CPAP side effect scale that is one of the few valid measures of the frequency and amount of CPAP side effects.
  1. A very large, All the time
  2. A large
  3. A moderate to large
  4. A moderate
  5. A small to moderate
  6. A small
  7. No, None, Not at all
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Self-Management
Number analyzed (Participants) | 90 | 100
units on a scale | 4.9 (1.04) | 5.1 (0.99)
Statistical Analysis 1: Comparison: Usual Care vs Self-Management; Test type: Superiority or Other; p = 0.96, t-test, 1 sided

6. Other Pre Specified Outcome: Quality of Well Being Scale (QWB-SA)
Description: The QWB-SA is a generic, preference-based measure that produces a single score appropriate for cost-effectiveness estimates and has been used in veteran and other general adult populations. The advantage of having a single, scaled score instead of multiple separate subscale domains is important for comparing interventions. The QWB-SA is a comprehensive measure of health-related quality of life that consists of 78-items and five sections: (I) acute and chronic symptoms; (II) self-care activities; (III) mobility; (IV) physical activity and performance of physical functioning; and (V) social activity. The level of functioning and the subjective symptom reports are then weighted by preference, or utility, on a scale that ranges from 0 (dead) to 1.0 (optimum function).
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Self-Management
Number analyzed (Participants) | 90 | 100
units on a scale | 0.56 (0.13) | 0.59 (014)
Statistical Analysis 1: Comparison: Usual Care vs Self-Management; Test type: Superiority or Other; p = 0.59, t-test, 1 sided

7. Other Pre Specified Outcome: Self-Efficacy
Description: Social-cognitive theory (SCT) measure
  1= Disagree Completely 5= Agree Completely 6= Not applicable
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Self-Management
Number analyzed (Participants) | 90 | 100
units on a scale | 3.9 (1.04) | 4.3 (0.8)
Statistical Analysis 1: Comparison: Usual Care vs Self-Management; Test type: Superiority or Other; p = 0.00, t-test, 1 sided

8. Other Pre Specified Outcome: Outcome Expectation
Description: Social-cognitive theory (SCT) measure
  1= Not at all important 5= Extremely important 6= Not applicable
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Self-Management
Number analyzed (Participants) | 90 | 100
units on a scale | 4.1 (0.9) | 4.5 (0.7)
Statistical Analysis 1: Comparison: Usual Care vs Self-Management; Test type: Superiority or Other; p = 0.02, t-test, 1 sided

9. Other Pre Specified Outcome: Center for Epidemiological Studies - Depression Scale (Short Form)
Description: The CES-D is a 10-item self-report measure of depression. The 10-item version has adequate predictive accuracy when compared to the original full-length 20-item version, as well as adequate test-retest correlations and discriminative validity.
  The total score is calculated by finding the sum of 10 items. Any score equal to or above 10 is considered depressed.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Self-Management
Number analyzed (Participants) | 90 | 100
units on a scale | 7.8 (5.9) | 7.2 (5.777)
Statistical Analysis 1: Comparison: Usual Care vs Self-Management; Test type: Superiority or Other; p = 0.08, t-test, 1 sided

10. Other Pre Specified Outcome: Epworth Sleepiness Scale (ESS)
Description: ESS is a widely used subjective measure of excessive daytime sleepiness in research and clinical settings. Participants are asked to indicate how likely they would be to fall asleep in eight different situations on a scale from 0 (not likely) to 3 (highly likely). The situations are designed to vary in sleep-inducing capacity. The ESS scoring range is 0-24, with higher scores reflecting greater daytime sleepiness.
Time Frame: 1 month
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Care | Self-Management
Number analyzed (Participants) | 90 | 100
units on a scale | 9.2 (4.8) | 8.1 (4.8)
Statistical Analysis 1: Comparison: Usual Care vs Self-Management; Test type: Superiority or Other; p = 0.38, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 1 month, 6 months, 1 year
Arm/Group | Usual Care | Self-Management
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/120
Other Adverse Events (participants affected / at risk) | 0/120 | 0/120

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes